CLINICAL TRIAL: NCT04801628
Title: Immediate Effects of TECAR Therapy on the Quadriceps Muscle Performance in Athlete
Brief Title: Immediate Effects of TECAR Therapy on the Quadriceps Muscle Performance in Athlete: A Randomized Crossover Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hamada Ahmed, Assistant Professor of Biomechanics and Ergonomics, Biomechanics Department, Faculty of Physical Therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: P.T.REC/012/003025
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: TECAR Therapy; Muscle Performance; Athletes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Tecar (Active Comparator): Transfer Electrode Capacitive and Resistive (TECAR) Therapy (radio frequency therapy; INDIBA, Spain) will be used. In CET mode, heat transfer is concentrated on the skin and superficial muscles, which are tissue with high electrolytes, while the RET mode focuses heat transfer on bones, tendons, joints, and deep muscles. In this study, both CET and RET modes will be applied to the participant' quadriceps for 15-20 minutes at stable frequency of 448 KHz. According to the manufacturer's guidelines for safety, the CET mode will be first implemented for 5 minutes. Then will be continued in RET mode using for the rest of the treatment. Participants will be asked to lie down comfortably, and treatment will be beginning.
  The intensity of the current will be set at the level of comfort between 0%-100%, averaging about 40%. TECAR therapy will be applied by a physical therapist for all participants.
  Interventions: Device: Active Tecar
- Placebo Tecar (Placebo Comparator): the same procedure as in active Tecar but the device not provide any radio frequency
  Interventions: Device: Placebo Tecar

INTERVENTIONS:
Device: Active Tecar — Active Tecar
  Arms: Active Tecar
Device: Placebo Tecar — Placebo Tecar
  Arms: Placebo Tecar

SUMMARY:
The experimental procedures will be composed of two sessions. The following steps will be constituted the first session: warm-up on the cycle ergometer, and familiarization with the isokinetic dynamometer then baseline measurement of isokinetic parameters. Afterward, the placebo or active TECAR therapy will be applied (according to the randomization). At the end, isokinetic parameters will be taken again. After 7 days, the second session will be performed following identical procedures to the first session. However, an inverse mode of TECAR therapy from the first session (placebo or active) will be applied for each individual. The two sessions will be held 7 days apart, either on a Sunday or Tuesday. Procedures are summarized in Figure 1. The dominant lower limb test will be used to elect the lower limb selected for isokinetic Dynamometer.

Figure 1: Timeline for the period of evaluation of groups (Active and Placebo TECAR).

Muscle performance measurement by Isokinetic Dynamometer:

The quadriceps muscles of dominant lower limb will be tested for all participants with Biodex isokinetic dynamometer (Biodex Medical System, Shiley, NY, USA, linked to IBM PC-computer software). Calibration of the Biodex for torque and angular speed will be done according to the prescribed manufacturer's guidelines before each recording session. Prior to assessment, the volunteers held a 5-min cycle ergometer warm up (speed in the range of 60-70 rpm and no load). After that, participants will be positioned with hip angle of 100o on the previously calibrated isokinetic dynamometer and will be properly aligned and stabilized with straps in order to avoid possible compensatory movements. Thus, the dominant knee axis (lateral epicondyle of the femur) of each subject was adjusted to the dynamometer rotation axis. The lever arm of the equipment was fixed approximately 2 cm above the tibial malleolus. The chair height, backrest distance, seat angle, and dynamometer base were adjusted for each subject and noted for the second session. Before starting the recording of isokinetic muscle performance, there will be a familiarization period with the apparatus consisting of five submaximal voluntary concentric muscle contractions in the full range of standardized and preprogrammed motion (90-20°) according to the guideline procedures of the dynamometer, with a constant angular velocity of 180°/s. the isokinetic protocol will be performed with a set of 60 concentric/eccentric contractions of quadriceps. The participants will be visually and verbally encouraged throughout the test protocol to achieve maximum effort from the beginning. The muscle performance, in terms of work fatigue index, peak torque, average power, and total work of the knee extensor muscles, will be evaluated by isokinetic dynamometry in accordance with the guidelines of the equipment manufacturer (Biodex Medical System Inc.).

Experimental protocol of TECAR therapy:

Immediately after the baseline measurement of muscle performance of each session, the participants will be received placebo or active TECAR therapy.

In this experiment, Transfer Electrode Capacitive and Resistive (TECAR) Therapy (radio frequency therapy; INDIBA, Spain) will be used. TECAR therapy is a systematic treatment for providing capacitive energy transfer (CET) and resistive energy transfer (RET). In CET mode, heat transfer is concentrated on the skin and superficial muscles, which are tissue with high electrolytes, while the RET mode focuses heat transfer on bones, tendons, joints, and deep muscles. In this study, both CET and RET modes will be applied to the participant' quadriceps for 15-20 minutes at stable frequency of 448 KHz. According to the manufacturer's guidelines for safety, the CET mode will be first implemented for 5 minutes. Then will be continued in RET mode using for the rest of the treatment. Participants will be asked to lie down comfortably, and treatment will be beginning.

The intensity of the current will be set at the level of comfort between 0%-100%, averaging about 40%. TECAR therapy will be applied by a physical therapist for all participants.

ELIGIBILITY:
Inclusion criteria

1. aged between 23 and 35 years.
2. body mass index of 20 to 25 kg/cm2
3. classified as irregularly active or active, who performed physical activity with a frequency of at least five times a week, totaling a minimum of 150 min per week, according to International Physical Activity Questionnaire (IPAQ)-Short Version and reports by participants were included.

Exclusion criteria

1. Those with previous musculoskeletal injury to the quadriceps femoris
2. Participants with hypersensitivity
3. A history of arthritis, injury, or surgery on the knee or hip
4. Participants that will be had a metal insert in the area requiring therapy were the excluded.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-12 (Estimated); Primary Completion 2021-03-12 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Peak torque of the quadriceps muscles of dominant lower limb will be tested for all participants with Biodex isokinetic dynamometer | 5 minutes from application of treatment
  The quadriceps muscles of dominant lower limb will be tested for all participants with Biodex isokinetic dynamometer
total work | 5 minutes from application of treatment
  The total work of quadriceps muscles of dominant lower limb will be tested for all participants with Biodex isokinetic dynamometer

SECONDARY OUTCOMES:
work fatigue index | 5 minutes from application of treatment
  The work fatigue index of quadriceps muscles of dominant lower limb will be tested for all participants with Biodex isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Hamada Ahmed, Cairo, Egypt